CLINICAL TRIAL: NCT01460381
Title: A Study to Investigate the Effect of CYP2C19 Phenotype on the Pharmacokinetics of LY2216684 in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Genotype on LY2216684
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14397; H9P-EW-LNDZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-03

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Quinidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2216684 + Quinidine (CYP2C19 poor metabolizers) (Experimental): Participants were predicted to have a cytochrome P450 (CYP)2C19 poor metabolizer (PM) phenotype, as determined by genotyping analysis.
  Period 1 (Days 1-7): a single, oral dose of 18 milligrams (mg) LY2216684 was administered on Day 1.
  Period 2 (Days 8-15): 300 mg quinidine sulfate controlled release was administered orally, once daily on Days 8-15. Additionally, a single, oral dose of 18 mg LY2216684 was administered on Day 11.
  Interventions: Drug: LY2216684; Drug: Quinidine
- LY2216684 (CYP2C19 extensive metabolizers) (Experimental): Participants were predicted to have a cytochrome P450 (CYP)2C19 extensive metabolizer (EM) phenotype, as determined by genotyping analysis.
  Period 1 (Days 1-7): a single, oral dose of 18 milligrams (mg) LY2216684 administered on Day 1.
  Period 2 (Days 8-15): EM participants did not participate in this period.
  Interventions: Drug: LY2216684

INTERVENTIONS:
Drug: LY2216684
Drug: Quinidine
  Other Names: Quinidine sulfate controlled release (CR)
  Arms: LY2216684 + Quinidine (CYP2C19 poor metabolizers)

SUMMARY:
The study will evaluate how genetic profiles respond to LY2216684 and the effect of Quinidine on the pharmacokinetics (PK) of LY2216684 in a specific genetic profile. Side effects will be documented.

DETAILED DESCRIPTION:
The human cytochrome P450 2C19 (CYP2C19) enzyme is a polymorphic enzyme yielding ultrarapid metabolizer, extensive metabolizer (EM), intermediate metabolizer, and poor metabolizer (PM) phenotypes. Enrollment in the study was limited to participants predicted to be CYP2C19 extensive metabolizers or CYP2C19 poor metabolizers, as determined by genotyping analysis.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Male participants: Agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug
* Female participants: Are women of child-bearing potential who test negative for pregnancy at the time of enrollment, have used a reliable method of birth control (not including hormonal contraceptives) for 4 weeks prior to administration of study drug, and agree to use a reliable method of birth control during the study and for 1 month following the last dose of the study drug or; Are women not of child-bearing potential due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation/occlusion) or menopause (at least 1 year without menses or 6 months without menses and a follicle stimulating hormone [FSH] level >40 milli-international units per milliliter [mIU/mL])
* Have a body weight >50 kilograms (kg)
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow for blood sampling as per the protocol
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the institutional review board (IRB) governing the site
* Have normal blood pressure (BP) and pulse rate (PR) (sitting position) as determined by the investigator
* Are predicted to have cytochrome P450 (CYP)2C19 extensive metabolizer (EM) or poor metabolizer (PM) phenotypes as determined by genotyping assessment
* Are predicted to have CYP2D6 EM phenotype as determined by genotyping assessment.

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies/intolerance to LY2216684 or quinidine, related compounds, or any components of the formulation
* Are persons who have previously received the investigational product in this study or have completed or withdrawn from this study or any other study investigating LY2216684 within 6 months prior to Screening.
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history or show evidence of significant active neuropsychiatric disease or have a history of suicide attempt or ideation
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Are women with a positive pregnancy test or women who are lactating
* Intend to use over-the-counter or prescription medication within 14 days prior to dosing or during the study unless deemed acceptable by the investigator and Sponsor's medical monitor. Exceptions include influenza vaccinations, the use of topical medication (provided there is no evidence of chronic dosing with the risk of systemic exposure), occasional use of acetaminophen/paracetamol/ibuprofen, and hormone replacement therapy including thyroid replacement (stable dose for at least 1 month).
* Have donated blood of more than 500 milliliters (mL) within the last month
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), or are unwilling to stop alcohol consumption 48 hours prior to dosing in Period 1 until Discharge (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study
* Consume 5 or more cups of coffee (or other beverages of comparable caffeine content) per day, on a habitual basis, or any participants unwilling to stop caffeine consumption from 48 hours prior to dosing in Period 1 until Discharge
* Have consumed grapefruit or grapefruit-containing products 30 days prior to enrollment or unwilling to abstain during the study
* Have a documented or suspected history of glaucoma
* Participants unwilling to adhere to the smoking restrictions of the Clinical Research Unit (CRU) while a resident of the CRU
* Use of known inhibitors and/or inducers of CYP2C19 and CYP2D6 (with the exception of quinidine per protocol) 30 days prior to enrollment or are unwilling to avoid them during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Period 1 (Days 1-7)
Arm/Group | LY2216684 + Quinidine (CYP2C19 Poor Metabolizers) | LY2216684 (CYP2C19 Extensive Metabolizers)
Started | 7 | 11
Received at Least 1 Dose of Study Drug | 7 | 11
Completed | 7 | 11
Not Completed | 0 | 0
Period: Period 2 (Days 8-15)
Arm/Group | LY2216684 + Quinidine (CYP2C19 Poor Metabolizers) | LY2216684 (CYP2C19 Extensive Metabolizers)
Started | 7 | 0 (CYP2C19 extensive metabolizers did not participate in Period 2.)
Completed | 6 (One participant was lost to follow-up after completing Period 2 and did not complete the study.) | 0 (CYP2C19 extensive metabolizers did not participate in Period 2)
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- LY2216684 + Quinidine (CYP2C19 Poor Metabolizers): Participants were predicted to have a cytochrome P450 (CYP)2C19 poor metabolizer (PM) phenotype, as determined by genotyping analysis.
  Period 1 (Days 1-7): a single, oral dose of 18 mg LY2216684 was administered on Day 1.
  Period 2 (Days 8-15): 300 mg quinidine sulfate controlled release was administered orally, once daily on Days 8-15. Additionally, a single, oral dose of 18 mg LY2216684 was administered on Day 11.
- LY2216684 (CYP2C19 Extensive Metabolizers): Participants were predicted to have a cytochrome P450 (CYP)2C19 extensive metabolizer (EM) phenotype, as determined by genotyping analysis.
  Period 1 (Days 1-7): a single, oral dose of 18 mg LY2216684 administered on Day 1.
  Period 2 (Days 8-15): EM participants did not participate in this period.
- Total: Total of all reporting groups
Arm/Group | LY2216684 + Quinidine (CYP2C19 Poor Metabolizers) | LY2216684 (CYP2C19 Extensive Metabolizers) | Total
Number analyzed (Participants) | 7 | 11 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (11.1) | 44.9 (12.1) | 43.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 9 | 10
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 2 | 9 | 11
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 11 | 18

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity [AUC(0-∞)] of LY2216684 in Cytochrome P450 (CYP)2C19 Extensive Metabolizers (EM) Versus Poor Metabolizers (PM)
Description: Blood samples were collected prior to and up to 120 hours following dosing of LY2216684 on Day 1 (Period 1) for the measurement of LY2216684 plasma concentrations.
Time Frame: Predose up to 120 hours post administration of LY2216684
Population: Participants who received at least 1 dose of LY2216684 and had evaluable LY2216684 plasma concentration data were included in the analysis. Participants who vomited within twice the median time to maximum observed drug concentration (tmax) following dosing of LY2216684 were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Groups:
- LY2216684 (CYP2C19 Poor Metabolizers): Participants were predicted to have a cytochrome P450 (CYP)2C19 poor metabolizer (PM) phenotype, as determined by genotyping analysis.
  Period 1 (Days 1-7): a single, oral dose of 18 mg LY2216684 was administered on Day 1.
- LY2216684 (CYP2C19 Extensive Metabolizers): Participants were predicted to have a cytochrome P450 (CYP)2C19 extensive metabolizer (EM) phenotype, as determined by genotyping analysis.
  Period 1 (Days 1-7): a single, oral dose of 18 mg LY2216684 administered on Day 1.
Arm/Group | LY2216684 (CYP2C19 Poor Metabolizers) | LY2216684 (CYP2C19 Extensive Metabolizers)
Number analyzed (Participants) | 7 | 7
nanograms*hours per milliliter (ng*h/mL) | 749 (37) | 698 (21)

2. Primary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) of LY2216684 in Cytochrome P450 (CYP)2C19 Extensive Metabolizers (EM) Versus Poor Metabolizers (PM)
Description: as for outcome 1
Time Frame: Predose up to 120 hours post administration of LY2216684
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | LY2216684 (CYP2C19 Poor Metabolizers) | LY2216684 (CYP2C19 Extensive Metabolizers)
Number analyzed (Participants) | 7 | 7
nanograms per milliliter (ng/mL) | 54.7 (28) | 54.8 (25)

3. Primary Outcome: Pharmacokinetics: Time to Maximum Observed Plasma Concentration (Tmax) of LY2216684 in Cytochrome P450 (CYP)2C19 Extensive Metabolizers (EM) Versus Poor Metabolizers (PM)
Description: as for outcome 1
Time Frame: Predose up to 120 hours post administration of LY2216684
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | LY2216684 (CYP2C19 Poor Metabolizers) | LY2216684 (CYP2C19 Extensive Metabolizers)
Number analyzed (Participants) | 7 | 7
hours | 2.00 [1.00 to 3.02] | 2.00 [1.92 to 5.00]

4. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity [(AUC(0-∞)] of LY2216684 + Quinidine in Cytochrome P450 (CYP)2C19 Poor Metabolizers (PM)
Description: Blood samples were collected prior to and up to 120 hours following coadministration of LY2216684 and quinidine on Day 11 (Period 2) for the measurement of LY2216684 plasma concentrations.
Time Frame: Predose up to 120 hours post administration of quinidine
Population: Participants who received at least 1 dose of LY2216684 and had evaluable LY2216684 plasma concentration data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Groups:
- LY2216684 + Quinidine (CYP2C19 Poor Metabolizers): Participants were predicted to have a cytochrome P450 (CYP)2C19 poor metabolizer (PM) phenotype, as determined by genotyping analysis.
  Period 2 (Days 8-15): 300 mg quinidine sulfate controlled release was administered orally, once daily on Days 8-15. Additionally, a single, oral dose of 18 mg LY2216684 was administered on Day 11.
Arm/Group | LY2216684 + Quinidine (CYP2C19 Poor Metabolizers)
Number analyzed (Participants) | 7
nanograms*hours per milliliter (ng*h/mL) | 1530 (34)

5. Secondary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) of LY2216684 + Quinidine in CYP2C19 Poor Metabolizers
Description: as for outcome 4
Time Frame: Predose up to 120 hours post administration of quinidine
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | LY2216684 + Quinidine (CYP2C19 Poor Metabolizers)
Number analyzed (Participants) | 7
nanograms per milliliter (ng/mL) | 66.9 (23)

6. Secondary Outcome: Pharmacokinetics: Time to Maximum Observed Plasma Concentration (Tmax) of LY2216684 + Quinidine in CYP2C19 Poor Metabolizers
Description: as for outcome 4
Time Frame: Predose up to 120 hours post administration of quinidine
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | LY2216684 + Quinidine (CYP2C19 Poor Metabolizers)
Number analyzed (Participants) | 7
hours | 3.00 [3.00 to 5.00]

ADVERSE EVENTS:
Groups:
- LY2216684 (CYP2C19 Extensive and Poor Metabolizers): Participants were predicted to have a cytochrome P450 (CYP)2C19 extensive metabolizer (EM) or poor metabolizer (PM) phenotype, as determined by genotyping analysis.
  Period 1 (Days 1-7): a single, oral dose of 18 milligrams (mg) LY2216684 administered on Day 1.
- Quinidine (CYP2C19 Poor Metabolizers): Participants were predicted to have a cytochrome P450 (CYP)2C19 poor metabolizer (PM) phenotype, as determined by genotyping analysis.
  Period 2 (Days 8-11, prior to LY2216684 dose): 300 mg quinidine sulfate controlled release was administered orally, once daily on Days 8-11.
- LY2216684 + Quinidine (CYP2C19 Poor Metabolizers): Participants were predicted to have a cytochrome P450 (CYP)2C19 poor metabolizer (PM) phenotype, as determined by genotyping analysis.
  Period 2 (Days 11-15, following LY2216684 dose): 300 mg quinidine sulfate controlled release was administered orally, once daily on Days 11-15. Additionally, a single, oral dose of 18 mg LY2216684 was administered on Day 11.
Arm/Group | LY2216684 (CYP2C19 Extensive and Poor Metabolizers) | Quinidine (CYP2C19 Poor Metabolizers) | LY2216684 + Quinidine (CYP2C19 Poor Metabolizers)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 10/18 | 1/7 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2216684 (CYP2C19 Extensive and Poor Metabolizers) (N=18) | Quinidine (CYP2C19 Poor Metabolizers) (N=7) | LY2216684 + Quinidine (CYP2C19 Poor Metabolizers) (N=7)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Social avoidant behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Testicular atrophy (Reproductive system and breast disorders) | 1/9 (1) | 0/5 (0) | 0/5 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days